CLINICAL TRIAL: NCT01223534
Title: Comparison of Two Strategies for Therapeutic Decision-making in Tuberculosis Contact Tracing: a Standard Strategy Based on Tuberculin Skin Test (TST) Alone vs TST Combined With QuantiFERON®-TB Gold In-Tube (QFT-IT)
Brief Title: QuantiFERON®-TB Gold In-Tube for the Diagnosis of Tuberculosis Infection in Contact Tracing Study.
Acronym: OPTIMIST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Cellestis (Industry)
Responsible Party: Principal Investigator, Miguel Santín Cerezales, PhD, MD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QFT-ECC-01; 2009-017430-49 (EudraCT Number); TRA-126 (Other Grant/Funding Number: Spanish Ministry of Health and Social Policy)
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Latent Tuberculosis Infection
Keywords: Tuberculosis; Latent tuberculosis infection; Tuberculin skin test; Interferon-gamma release assays; Contact-tracing study
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A, Standard practice, TST (Active Comparator): Participants allocated to screening as stablished by current practice (TST)
  Interventions: Drug: Preventive treatment with Isoniazid.
- Arm B, Experimental, TST plus QFT-IT (Experimental): Participants allocated to screening with TST, and if positive, followed by QFT-IT to confirm tuberculosis infection.
  Interventions: Drug: Preventive treatment with Isoniazid

INTERVENTIONS:
Drug: Preventive treatment with Isoniazid. — If TST positive: participant will be treated with Isoniazid 300 mg/d, for 6 months.
  Arms: Arm A, Standard practice, TST
Drug: Preventive treatment with Isoniazid — If QFT-IT positive, Isoniazid 300 mg/d, for 6 months.
  Arms: Arm B, Experimental, TST plus QFT-IT

SUMMARY:
Hypothesis: a combined strategy of tuberculin skin test (TST) followed by QuantiFERON-TB Gold In-Tube (QFT-IT) to confirm positivity (tuberculosis infection,in contact-tracing study will allow avoiding unnecessary preventive treatment without increasing rates of tuberculosis cases among contacts screened.

Aim of the study: to compare a combined strategy of the TST and the QFT-IT with TST alone for the diagnosis of tuberculosis infection and for therapeutic decision in contact tracing study.

Design and setting: Prospective, multicentre, comparative study in 12 hospitals in Spain.

Study population: 870 subjects, household contacts of patients with culture positive pulmonary and/or laryngeal tuberculosis will be randomized to one of two strategies: Arm A (standard practice), in which treatment decisions will be based on the TST result, and Arm B (experimental), in which treatment decisions will be based on the QFT result.

Interventions: participants in arm A will undergo TST; participants in arm B will undergo TST, and, in case of a positive result, QFT-IT as well. Participants with positive TST (arm A) and positive QFT-IT (arm B) will be diagnosed with tuberculosis infection and will be treated with isoniazid for 6 months. All participants will be followed for two years.

End-points of evaluation: development of tuberculosis and proportion of subjects for whom treatment is prescribed in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Close contact of a pulmonary and/or laryngeal tuberculosis case.
* Written informed consent.

Exclusion Criteria:

* HIV infection.
* Immunosuppression other than HIV, such as decompensated liver disease, chronic renal failure, corticosteroids treatment, malignancy under chemotherapy therapy.
* Prior tuberculosis or positive TST.
* Strain resistant to Isoniazid (index case).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 871 (Actual)
Dates: Start 2010-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Development of tuberculosis. | Assessment of primary end-point: 24 months after randomization.

SECONDARY OUTCOMES:
Prescription of treatment. | The day 0 (visit 2) after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Santin, MD, Study Director — Bellvitge University Hospital, Bellvitge Institute for Biomedical Research (IDIBELL)
Locations (1):
- Bellvitge University Hospital, IDIBELL, L'Hospitalet de Llobregat, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munoz L, Santin M, Alcaide F, Ruiz-Serrano MJ, Gijon P, Bermudez E, Dominguez-Castellano A, Navarro MD, Ramirez E, Perez-Escolano E, Lopez-Prieto MD, Gutierrez-Rodriguez J, Anibarro L, Calvino L, Trigo M, Cifuentes C, Garcia-Gasalla M, Payeras A, Gasch O, Espasa M, Aguero R, Ferrer D, Casas X, Gonzalez-Cuevas A, Garcia-Zamalloa A, Bikuna E, Lecuona M, Galindo R, Ramirez-Lapausa M, Carrillo R; OPTIMIST Study Team. QuantiFERON-TB Gold In-Tube as a Confirmatory Test for Tuberculin Skin Test in Tuberculosis Contact Tracing: A Noninferiority Clinical Trial. Clin Infect Dis. 2018 Jan 18;66(3):396-403. doi: 10.1093/cid/cix745. PMID 29020191